CLINICAL TRIAL: NCT02818738
Title: A Multicenter, Randomised, Double-blind Placebo-controlled Trial Assessing the Efficiency of Levamisole for Maintaining Remission After the First Flare of Steroid Sensitive Nephrotic Syndrome in Children.
Brief Title: Efficiency of Levamisole for Maintaining Remission After the First Flare of Steroid Sensitive Nephrotic Syndrome in Children
Acronym: NEPHROVIR3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150904
Record Dates: First submitted 2016-06-08; First posted 2016-06-30 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: First Manifestation of Steroid Sensitive Nephrotic Syndrome
Keywords: Idiopathic nephrotic syndrome; Steroid sensitive nephrotic syndrome; Levamisole; Prednisone; Children
MeSH Terms: conditions — Nephrosis, Lipoid; Nephrotic Syndrome | interventions — Levamisole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levamisole Hydrochloride (Experimental): Dosage : 5, 10, 25 et 50mg. Dosage form : oral tablets, coated and non dividable for taste-masking Posology : 2.5 mg/kg on alternate days maximum 150mg. Treatment duration : 6 months
  Interventions: Drug: Levamisole Hydrochloride
- Placebo (Placebo Comparator): matching verum
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levamisole Hydrochloride — Dosage : 5, 10, 25 et 50 mg. Dosage form : oral tablets, coated and non dividable for taste-masking Posology : 2.5 mg/kg on alternate days maximum 150mg. Treatment duration : 6 months
  Arms: Levamisole Hydrochloride
Other: Placebo — matching verum
  Arms: Placebo

SUMMARY:
Idiopathic Nephrotic Syndrome is sensitive to steroid in 90% of children. However, most patients relapse and become steroid-dependant, with a long lasting relapsing course. The aim of this study is to assess the efficiency of a 6-months levamisole course, given early after first remission, on maintaining a relapse-free course at 12 months.

DETAILED DESCRIPTION:
Introduction (INS) is likely a primal immune disorder. Initial treatment relies on steroid therapy. NS is sensitive to steroid in more than 90% of cases, with an excellent renal prognosis. Nevertheless, 80% of patients with steroid sensitive NS do relapse, 60% within the first year. 2/3 of them will experience steroid dependency, with a long lasting relapsing course. These patients require further immunosuppressive drugs as steroid sparing agents, such as mycophenolate, cyclophosphamide, calcineurin inhibitors or rituximab. Morbidity is high and related both to the duration of the disease, sometimes until adulthood, and to treatments side effects.

Levamisole is an immunomodulator that has been used for more than thirty years in the treatment of steroid-dependent or frequently relapsing NS. Its major advantages are its immunomodulatory action and lower and reversible toxicity.

Exact physiopathology of both INS and levamisole action remain unknown. Nevertheless, we make the hypothesis that very early treatment with levamisole may enhance its efficiency and modify the disease's course.

This is the first trial to assess the efficiency of levamisole in increasing duration of remission after the first manifestation of INS.

Design :

* A multicenter, double-blind, placebo-controlled, randomised clinical trial.
* 38 centers participate to the recruitment : 3 Pediatric Nephrology units and 35 General Pediatric units.
* 20 centers participate to the randomized phase.

Sample size :

156 patients, 78 in each group

Treatment groups :

1. Levamisole Hydrochloride Dosage : 5, 10, 25 et 50mg. Dosage form : oral tablets Posology : 2.5 mg/kg on alternate days maximum 150mg. Treatment duration : 6 months
2. placebo : matching verum

Assessment :

Study visits at inclusion, M1 (randomisation), M3, M6, M9, M12. Supplementary visit if relapse occurs.

Statistical procedure Analysis of efficiency will be performed on intention to treat population. Analysis of tolerance will be performed on randomized patients who have received at least one dose of treatment.

No intermediary analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age 24 months < age < 16 years
* Diagnosis of first manifestation of INS defined by:
* hypoalbuminemia < 25g/l, proteinuria > 0.20 g/mmol of urinary creatinine
* normal C3 fraction of complement
* Use of mechanical contraception for patients of reproductive age throughout the research period
* Beneficiary of a social protection scheme (except AME)
* Written informed consent from one of both parents
* Ability to realise follow-up in full

Exclusion Criteria:

* Anteriority of INS
* Pregnancy, breast feeding or planned pregnancy during the study
* Malignant pathology (antecedent or ongoing), diabetes, liver disease
* Hypersensitivity to levamisole or its excipients (lactose)

Ages: 24 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients still in remission at 12 months after first flare of INS. | 12 months
  number of patients who did not relapse compared to the number of patients who had relapsed after first flare of INS.

SECONDARY OUTCOMES:
Compare within levamisole and placebo groups the duration of remission. | first relapse
  number of days between the first flare and first relapse or up to the corticodependence level in the event of relapse in the course of decreasing corticosteroid therapy.
Compare within levamisole and placebo groups the frequency and level of steroid dependency | 12 months
  Proportion of corticodependent patients and level of steroid dependency
Compare within levamisole and placebo groups the treatment tolerance | 12 months
  Frequency of adverse events apparition and frequency of discontinuation of treatment secondary at a adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Claire DOSSIER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526